CLINICAL TRIAL: NCT01752049
Title: Topical Anti-angiogenic Therapy for Telangiectasia in HHT: Proof of Concept
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of California, San Francisco (Other); The Hospital for Sick Children (Other); University of Toronto (Other); Sunnybrook Health Sciences Centre (Other); Toronto Metropolitan University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVMC 6207; 2U54NS065705-06 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: Hereditary Hemorrhagic Telangiectasia; Anti-angiogenic Therapy; vascular malformations; HHT
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Vascular Malformations | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical timolol maleate (Active Comparator): Drug: • Topical timolol maleate 0.5% drops
  * Topical timolol maleate 0.5% drops
  * Applied twice daily for 12 weeks (84 days) or until disappearance of lesions
  * Study drops will be applied to 3 cutaneous telangiectasias per patient telangiectasia per patient).
  Interventions: Drug: Topical timolol maleate
- Placebo (Placebo Comparator): placebo saline drops
  -Applied twice daily for 12 weeks (84 days) or until disappearance of lesions to one cutaneous telangiectasias per patient.
  Interventions: Drug: placebo saline drops

INTERVENTIONS:
Drug: Topical timolol maleate — * Topical timolol maleate 0.5% drops
  * Applied twice daily for 12 weeks (84 days) or until disappearance of lesions
  * Study drops will be applied to 3 cutaneous telangiectasias per patient
  Other Names: Topical timolol maleate 0.5% drops
  Arms: Topical timolol maleate
Drug: placebo saline drops — Applied twice daily for 12 weeks (84 days) or until disappearance of lesions to 1 cutaneous telangiectasias per patient.
  Arms: Placebo

SUMMARY:
Hereditary hemorrhagic telangiectasia (HHT) is a hereditary vascular condition characterized by the development of abnormal connections between arteries and veins throughout the body, called vascular malformations. These abnormal blood vessels are referred to as arteriovenous malformations (AVM) if they are large and telangiectasias if they are small. Telangiectasias develop due to irregular growth of blood vessels.

Anti-angiogenic therapy, such as the drug Apo-Timop, curbs the growth of new blood vessels. Apo-Timop is included in a class of medications called beta-blockers. Anti-angiogenic therapies exert their beneficial effects in a number of ways: by disabling the agents that activate and promote cell growth, or by directly blocking the growing blood vessel cells.

The investigators think that anti-angiogenic therapy may lead to the shrinking of telangiectasia in people with HHT. The investigators hope that this study will provide us with proof of this concept and might lead to the development and study of anti-angiogenic therapies to help improve the lives of individuals with vascular malformations.

DETAILED DESCRIPTION:
This is a small study of 5 patients from St. Michael's Hospital who have HHT and at least 5 typical telangiectasias.

Patients who anticipate a major surgery during this study or are pregnant, breast feeding or on other beta blocker medication may not enroll in this study.

This study lasts 12 weeks (84 days). During this time, subjects will apply a drop of either Apo-timop 0.5% or a placebo solution to 4 telangiectasias twice daily.

The active study medication is called Apo-Timop and is a clear liquid solution stored in a bottle. An eye dropper is used for application.

* Apo-timop will be applied to 3 telangiectasias and
* a placebo will be applied to one telangiectasia A placebo is an inactive substance, with no active medication in it, and it looks the same as the real medication. There is no potential harm of receiving the placebo. It is necessary to use a placebo to make sure that the effect of Apo-timop can be determined without any bias.

Subjects will receive four numbered bottles for every 28 day period as well as a photo which indicates which bottle is to be applied to which telangiectasia.

Neither the subject nor the research staff will know which telangiectasia will receive the placebo.

Apo-timop, is not part of the standard therapeutic regimen for HHT. It is a Health Canada approved medication which is applied as an eye drop, that has been shown to reduce pressure in the eye and is commonly used for glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Definite clinical or genetic diagnosis of HHT
2. Known ENG or ALK1 mutation (personal or familial)
3. Age>=18 years
4. At least 5 typical (round/ovoid, not spider or linear) cutaneous telangiectasia (size range 2-5mm) on hands (not including lesions on over inter-phalangeal joints) or face

Exclusion Criteria:

1. Contraindication to systemic beta-blocker (severe asthma, severe COPD, sinus bradycardia, 2nd or 3rd degree AV block, overt heart failure, hypotension, allergy/intolerance/ hypersensitivity to timolol)
2. Current treatment with systemic beta-blocker
3. Current participation in other therapeutic trial for HHT
4. Current pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Faughnan, MD MSc FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each Participant received both treatment and placebo
Units Other Than Participants: Telangiectasia (Lesions)
Groups:
- Topical Timolol Maleate: Topical timolol maleate 0.5% drops will be applied twice daily for 12 weeks (84 days) or until disappearance of lesions on 3 cutaneous telangiectasias per patient (total of 5 patients)
- Placebo: placebo saline drops will be applied twice daily for 12 weeks (84 days) or until disappearance of lesions to one cutaneous telangiectasias per patient (same 5 patient as Topical treatment group)
Period: Overall Study
Arm/Group | Topical Timolol Maleate | Placebo
Started | 5; 15 Telangiectasia (Lesions) | 5; 5 Telangiectasia (Lesions)
Completed | 5; 15 Telangiectasia (Lesions) | 5; 5 Telangiectasia (Lesions)
Not Completed | 0; 0 Telangiectasia (Lesions) | 0; 0 Telangiectasia (Lesions)

BASELINE CHARACTERISTICS:
Population: Total 5 participants treated (15 treatment lesions and 5 placebo lesions)
Groups:
- All Study Participants: Drug: • Topical timolol maleate 0.5% drops
  * Topical timolol maleate 0.5% drops
  * Applied twice daily for 12 weeks (84 days) or until disappearance of lesions
  * Study drops will be applied to 3 cutaneous telangiectasias per patient telangiectasia per patient).
  Topical timolol maleate: • Topical timolol maleate 0.5% drops
  * Applied twice daily for 12 weeks (84 days) or until disappearance of lesions
  * Study drops will be applied to 4 cutaneous telangiectasias per patient (timolol drops for 3 telangiectasia per patient and placebo drops to 1 telangiectasia per patient).
Arm/Group | All Study Participants
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Area of Treated Telangiectasia.
Description: Change in lesion area (compared with baseline measurement) of treated telangiectasia.
Time Frame: 84 days
Population: 5 participants enrolled, each participant have Hereditary Hemorrhagic Telangiectasia (HHT) and have at least 5 typical telangiectasias on their hands or face.
Measure: Geometric Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesion (Telangiectasia)
Groups:
- Topical Timolol Maleate: 5 Participants received Topical timolol maleate 0.5% drops. Applied twice daily for 12 weeks (84 days) or until disappearance of lesions Study drops will be applied to 3 cutaneous telangiectasias per patient
- Placebo: The same 5 participants will receive placebo saline drops on one cutaneous telangiectasia. Applied twice daily for 12 weeks (84 days) or until disappearance of lesions to one cutaneous telangiectasias per patient.
Arm/Group | Topical Timolol Maleate | Placebo
Number analyzed (Participants) | 5 | 5
Number analyzed (Lesion (Telangiectasia)) | 15 | 5
mm^2 | -6 (11) | -8 (17)

2. Secondary Outcome: Descriptive Changes in Histopathology in Baseline vs Treated Lesions
Time Frame: 84 days
Population: No data collected
Arm/Group | Topical Timolol Maleate | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Serum Angiogenic Markers
Time Frame: 84 days
Population: No data collected
Arm/Group | Topical Timolol Maleate | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Stability of Area of Untreated Telangiectasias Over the 84 Day Period
Time Frame: 84 days
Population: No data collected
Arm/Group | Topical Timolol Maleate | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Blood Flow Velocity and Volume Flow Rates
Time Frame: 84 days
Population: No data collected
Arm/Group | Topical Timolol Maleate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 84 days
Groups:
- Topical Timolol Maleate: 5 patients received Topical timolol maleate 0.5% drops. Applied twice daily for 12 weeks (84 days) Study drops were applied to 3 cutaneous telangiectasias per patient. Each patient had 2 lesional biopsies (one at baseline, and one at end of treatment)
- Placebo: The same 5 patients received placebo saline drops for one telangiectasia each. The placebo drops were applied twice daily for 12 weeks (84 days)
Arm/Group | Topical Timolol Maleate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Timolol Maleate (N=5) | Placebo (N=5)
Minor infection at biopsy site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — expected adverse event -Biopsy site
Minor bleeding at biopsy site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — expected adverse event -Biopsy site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT01752049/Prot_SAP_000.pdf